CLINICAL TRIAL: NCT03275233
Title: Psychiatric Comorbidities in Patient With Painful Peripheral Neuropathy
Brief Title: Psychiatric Comorbidities in Patients With Painful Peripheral Neuropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Andrew Ibrahim Farag, Principal Investigator, Assiut University
Other Study IDs: PCIPWPPN
Record Dates: First submitted 2017-08-29; First posted 2017-09-07 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-01

CONDITIONS: Painful Peripheral Neuropathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Psychiatric comorbidities in patient with Painful Peripheral neuropathy

DETAILED DESCRIPTION:
Neuropathic pain has been redefined by the International Association for the Study of Pain, as'' pain caused by a lesion or disease of somatosensory system''.Diabetic peripheral neuropathy is the result of nerve damage in the toes, feet, and hands . Approximately 50% of those diabetic peripheral neuropathy have neuropathic pain .

Patients with persistent neuropathic pain experience work disability and activity limitation, with a substantial impact on their social functioning. As any chronic pain state comorbid depression, anxiety and sleep disturbance are common occurring in up to one half of those with painful neuropathy.

The relationship between chronic pain and cognitive function has not been adequately studied and little is known about cognitive functioning in neuropathic conditions. This may be because the clinicians pay more attention to psychiatric comorbidities, such as depression and anxiety.Although chronic pain associated with cognitive deficits may impact on everyday behaviour and interfere with emotional decision-making tasks.

In a cross-sectional survey at the Mayo clinic, the prevalence of clinician-diagnosed symptomatic or painful diabetic peripheral neuropathy was 13-15% out of 78% of those with any type of diabetic peripheral neuropathy . Many patients with diabetic peripheral neuropathy experience neuropathic pain, typically characterized as burning, electric, sharp and shooting which initially starts in both feet and may progress to involve calves, fingers, and hands (stocking and glove pattern) .

Recently it has been demonstrated an association between diabetes , diabetes complication and impairment of mental health and particular emphasis has been placed on the association between painful diabetic sensory neuropathy with depression .

ELIGIBILITY:
Inclusion Criteria:

1. Any female or male diabetic patient is aged 18 years or above had diabetic peripheral neuropathy.
2. patients must be able to swallow tables

Exclusion Criteria:

1. Patients have other comorbid psychiatric disorders or psychological troubles that is not secondary to diabetic neuropathy according to clinical and psychiatric evaluation,
2. Patients have any other causes of pain condition, or had skin conditions that are likely to confound the assessment of diabetic peripheral neuropathic pain.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with painful peripheral neuropathy
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-09-04 (Estimated); Primary Completion 2020-01-04 (Estimated); Study Completion 2021-01-04 (Estimated)

PRIMARY OUTCOMES:
Psychiatric comorbidities in diabetic patients with painful(symptomatic)peripheral neuropathy. | 6 month
  1- Pain assessment using visual analogue scale (VAS).

IPD SHARING:
Plan to Share IPD: Undecided